CLINICAL TRIAL: NCT00411957
Title: The Pharmacokinetics of Atazanavir / Ritonavir 200/100 OD Versus 300/100 mg OD in Combination With 2 NRTIs in HIV Pre-treated Patients
Brief Title: Pharmacokinetic Study of 2 Doses of ATV/r OD + 2 NRTIs in Thai HIV-1 Infected Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 073
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: atazanavir/ritonavir; pharmacokinetic of ATV/r200/100 OD+2NRTIs
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): ATV/r 300/100 mg
  Interventions: Drug: Atazanavir
- 2 (Active Comparator): ATV/r 200/100 mg OD
  Interventions: Drug: Atazanavir

INTERVENTIONS:
Drug: Atazanavir — ATV/r 300/100mg OD vs ATV/r 200/100 mg OD

SUMMARY:
Several studies from HIV-NAT have demonstrated high nevirapine, indinavir, saquinavir and lopinavir/r levels when compared to Caucasian patients. Until now, the pharmacokinetics of atazanavir have not been explored in a Thai population. We postulate that ATV levels, as with other PIs, are higher in Thai people. Therefore, the level of ATV in ATV/RTV 300/100 OD may be higher than the acceptable range and could be associated with ATV related toxicity.

DETAILED DESCRIPTION:
We are interested in once daily ATV/RTV 200/100 mg OD because of the convenience, reduction in ATV doses which may improve adherence while reducing toxicity and cost. There are limited prospective studies evaluating pharmacokinetic and long term efficacy and safety of atazanavir/ritonavir once daily dose in combination of NRTIs in HIV-1 pretreated patients. We believe that the PK parameters of ATV/RTV given at 200/100mg daily in Thai patients will be equivalent to the ATV/RTV 300/100mg once daily dosing in Caucasian patients when combined with 2NRTIs, and that the once daily regimen will have better safety, tolerability profile, and cost saving while maintaining good CD4 and VL outcome. If, the pharmacokinetic profile of ATV/RTV 200/100 mg OD + 2NRTIs is in acceptable range or comparable with standard dose of ATV/RTV 300/100 mg OD, long term efficacy will be explored later.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adults HIV patients currently using ATV/RTV 300/100 mg OD plus 2 NRTIs
* HIV RNA < 50 copies/ml

Exclusion Criteria:

* Inability to understand the nature and extent of the study and the procedures required.
* ALT/ AST more than 5x upper limit
* Relevant history or current condition, illness that might interfere with drug absorption, distribution, metabolism or excretion.
* Use of concomitant medication that may interfere with the pharmacokinetics of atazanavir, and ritonavir
* History of sensitivity/idiosyncrasy to the drug or chemically related compounds which may be employed in the study.
* Active drug abuse or heavy alcoholic drinking
* History of sensitivity/idiosyncrasy to the drug or chemically related compounds which may be employed in the study.
* Active drug abuse or heavy alcoholic drinking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
the pharmacokinetics of atazanavir/ritonavir (ATV/RTV) 200/100 mg once daily in a sample of 22 patients experiencing virological success | 1 year

SECONDARY OUTCOMES:
The pharmacokinetic and pharmacodynamic between these patients and data from Thai cohort treated with ATV/RTV 300/100 mg OD | 4 weeks
short term safety, tolerability and efficacy data in these PK participating patients | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — HIV-NAT Thai Red Cross AIDS Research Center
Locations (1):
- HIV-NAT, Thai Red Cross AIDS Research Center, Bangkok, Thailand

REFERENCES:
- [Result] Avihingsanon A, van der Lugt J, Kerr SJ, Gorowara M, Chanmano S, Ohata P, Lange J, Cooper DA, Phanuphak P, Burger DM, Ruxrungtham K. A low dose of ritonavir-boosted atazanavir provides adequate pharmacokinetic parameters in HIV-1-infected Thai adults. Clin Pharmacol Ther. 2009 Apr;85(4):402-8. doi: 10.1038/clpt.2008.244. Epub 2008 Dec 31. PMID 19118378
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org